CLINICAL TRIAL: NCT06984653
Title: Evaluation of the Effect of Scalp Block on Bispectral Index Values During Skull Pinning; Prospective Observational Study
Brief Title: Effect of Scalp Block on Bispectral Index Values During Skull Pinning
Status: Completed | Type: Observational
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Halide Hande Şahinkaya, MD, Bozyaka Training and Research Hospital
Other Study IDs: scalp block
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-08

CONDITIONS: Bispectral Index
Keywords: bispectral index; skull pinning; craniotomy; scalp block

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group S: Group of patients who will be performed scalp block
- Group LA: Group of patients who will be performed local anesthetic infiltration into pin sites

SUMMARY:
The aim of this prospective observational study is to evaluate the scalp block on bispectral index (BIS) values during skull pinning in patients undergoing craniotomy. The main questions it aims to answer are;

1. Is there an increase in BIS during skull pin insertion when scalp block is performed?
2. Are there any hemodynamic changes during skull pin insertion when scalp block is performed? Participants will be observed for BIS values and hemodynamic changes during skull pinning.

DETAILED DESCRIPTION:
In neurosurgery, maintaining arterial blood pressure within normal limits and keeping the depth of anesthesia under control constitute the basis of anesthesia management in patients undergoing craniotomy. Sudden hemodynamic changes due to inadequate analgesia and depth of anesthesia result in increased intracranial pressure. As a result of increased intracranial pressure, conditions such as hemorrhage and herniation may be encountered in the brain with decreased compliancy due to intracranial space-occupying mass.

Bispectral index (BIS) is a monitoring technique that evaluates the depth of anesthesia and allows optimal anesthetic agent administration. With the help of a sensor placed on the patient's forehead, electroencephalography (EEG) waves are analyzed and converted into numerical data by the processor. The incidence of anesthesia awareness decreases in general anesthesia applications with a BIS value below 60.

Tachycardia and hypertension may develop despite adequate depth of anesthesia with nociculus stimulation at the skin incision during placement of the skull pins. This is especially undesirable in patients with hypertension. Local anesthetic infiltration can be applied to the pin sites or the sensory innervation of the skin can be blocked by scalp block. Previous studies have shown positive effects of local anesthetic infiltration on BIS values during skull pinning.

The primary aim of our study is to evaluate the effect of scalp block on BIS values during skull pin insertion. Secondary aim is to evaluate the hemodynamic changes. The changes will be statistically analyzed between those who will be administered scalp block and those who will not.

The study is planned as a prospective cross-sectional observational study. Patients over 18 years with ASA (American Society of Anesthesiology) score I-II-III who will undergo elective craniotomy for supratentorial mass excision will be included in the study. They will be recorded in two groups as Group S (scalp block) and Group LA (local anesthesia). Scalp block or local anesthetic infiltration will be the choice of the anesthesiologist who is independent of the study and cares for the patient. There will be no intervention in anesthetic applications.

Systolic, diastolic and mean arterial blood pressure, heart rate and bispectral index values before and at 1, 3, 5, 10 and 15 minutes after skull pinnig will be recorded from anesthesia observation form.

Parametric descriptive values will be given as mean and standard deviation, and non-parametric values will be given as n (%) and median and IQR (interquartile range). The conformity of the data to normal distribution will be evaluated by one sample Kolmogorov-Smirnov test. Comparisons of quantitative data conforming to normal distribution will be made with Student T test and comparisons of data not conforming to normal distribution will be made with Mann Whitney U test. Chi-Square test will be used to compare qualitative data. For the analyses, the significance level will be accepted as p<0.05 at 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective craniotomy for supratentorial mass excision
* Above 18 years of age
* ASA score I-II-III

Exclusion Criteria:

* Patients without written approval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective craniotomy for supratentorial mass excision
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2025-05-25 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Bispectral index period 1 | Just before skull pinning
  Bispectral index value will be noted through BIS monitoring via the BIS sensor attached to the frontal area. BIS index is a numerical scale between 0 and 100, where 100 is completely awake and 0 is isoelectric status. BIS value between 40-60 shows the adequate depth of anesthesia.
Bispectral index period 2 | 1 minute after skull pinning
  BIS values between 40-60 show the adequate depth of anesthesia.
Bispectral index period 3 | 3 minutes after skull pinning
  BIS values between 40-60 show the adequate depth of anesthesia.
Bispectral index period 4 | 5 minutes after skull pinning
  BIS values between 40-60 show the adequate depth of anesthesia.
Bispectral index period 5 | 10 minutes after skull pinning
  BIS values between 40-60 show the adequate depth of anesthesia.
Bispectral index period 6 | 15 minutes after skull pinning
  BIS values between 40-60 show the adequate depth of anesthesia.

SECONDARY OUTCOMES:
systolic blood pressure 1 | Just before skull pinning
diastolic blood pressure 1 | Just before skull pinning
mean blood pressure 1 | Just before skull pinning
Heart rate 1 | Just before skull pinning
systolic blood pressure 2 | 1 minute after skull pinning
diastolic blood pressure 2 | 1 minute after skull pinning
mean blood pressure 2 | 1 minute after skull pinning
Heart rate 2 | 1 minute after skull pinning
systolic blood pressure 3 | 3 minutes after skull pinning
diastolic blood pressure 3 | 3 minutes after skull pinning
mean blood pressure 3 | 3 minutes after skull pinning
heart rate 3 | 3 minutes after skull pinning
systolic blood pressure 4 | 5 minutes after skull pinning
diastolic blood pressure 4 | 5 minutes after skull pinning
mean blood pressure 4 | 5 minutes after skull pinning
heart rate 4 | 5 minutes after skull pinning
systolic blood pressure 5 | 10 minutes after skull pinning
diastolic blood pressure 5 | 10 minutes after skull pinning
mean blood pressure 5 | 10 minutes after skull pinning
heart rate 5 | 10 minutes after skull pinning
systolic blood pressure 6 | 15 minutes after skull pinning
diastolic blood pressure 6 | 15 minutes after skull pinning
mean blood pressure 6 | 15 minutes after skull pinning
heart rate 6 | 15 minutes after skull pinning

CONTACTS AND LOCATIONS:
Overall Officials: Halide Hande ŞAHİNKAYA, MD, Principal Investigator — Izmir City Hospital; Gözde Gürsoy Çirkinoğlu, MD, Study Chair — Izmir City Hospital; Cafer Ak, MD, Study Chair — Izmir City Hospital; Sermin Altunbaş, MD, Study Chair — Izmir City Hospital; Zeki Tuncel Tekgül, Professor, Study Chair — Izmir City Hospital
Locations (1):
- Izmir City Hospital, Izmir, Turkey (Türkiye)